CLINICAL TRIAL: NCT05615623
Title: A Safety and Feasibility Study to Evaluate Blood Brain Barrier Disruption Using Exablate MR Guided Focused Ultrasound in Combination With Doxorubicin in Treating Pediatric Patients With Diffuse Intrinsic Pontine Gliomas (DIPG)
Brief Title: Blood Brain Barrier (BBB) Disruption Using Exablate Focused Ultrasound With Doxorubicin for Treatment of Pediatric DIPG
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: InSightec (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: BT016C
Record Dates: First submitted 2022-11-07; First posted 2022-11-14 (Actual); Last update posted 2025-04-30 (Actual); Status verified 2025-04

CONDITIONS: Brain Tumor
Keywords: DIPG; Focused Utrasound; Chemotherapy; Phase I trial; Pediatrics
MeSH Terms: conditions — Brain Neoplasms | interventions — Doxorubicin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Blood Brain Barrier Disruption (BBBD) (Experimental): Exablate MR Guided Focused Ultrasound for Blood Brain Barrier Disruption with Doxorubicin for treating pediatric patients with DIPG
  Interventions: Device: Exablate; Drug: Doxorubicin

INTERVENTIONS:
Device: Exablate — Blood Brain Barrier Disruption (BBBD) via Exablate Type 2 system with microbubble resonators on the day of Doxorubicin infusion to treat DIPG brain tumors
  Other Names: Exablate BBBD
Drug: Doxorubicin — Doxorubicin infusion
  Other Names: Adriamycin; Rubex

SUMMARY:
The purpose of this study is to evaluate the safety and efficacy of targeted blood brain barrier disruption with Exablate Model 4000 Type 2.0/2.1 in combination with Doxorubicin therapy for the treatment of DIPG in pediatric patients

DETAILED DESCRIPTION:
This is a prospective, single arm, non-randomized feasibility study to evaluate the safety, feasibility and preliminary efficacy of Blood Brain Barrier Disruption (BBBD) using the Exablate Type 2 system in pediatric patients with Diffuse Intrinsic Pontine Gliomas (DIPG) undergoing Doxorubicin chemotherapy. The study will be conducted at a single center in Canada. Patients will undergo 3 treatment cycles, approximately 4 -6 weeks apart. The study aims to establish feasibility and safety of Exablate BBBD in conjunction with Doxorubicin in the treatment of pediatric DIPG and assess preliminary efficacy in this patient population.

ELIGIBILITY:
Inclusion Criteria:

* Age between 5 and 18 years, inclusive
* Patient diagnosed with DIPG
* At least 4-week and not greater than 12 weeks from completion of radiation therapy
* Post-radiation imaging does not show evidence of necrosis/ hemorrhage or other features that contraindicate MRgFUS
* Able to attend all study visits and with life expectancy of at least 6 months
* Able and willing to give consent and/or assent or have a legal guardian who is able and willing to do so
* If on steroids, stable or decreasing dose for at least 7 days prior to study entry
* If brain surgery occurred, at least 14 days passed since last brain surgery and the patient is fully recovered and neurologically stable

Exclusion Criteria:

* Evidence of cranial or systemic infection
* Known life-threatening systemic disease
* Previous treatment with complete cumulative doses of Doxorubicin, daunorubicin, idarubicin, and/or other anthracyclines and anthracenediones
* Contraindication to Doxorubicin. - Known sensitivity to DEFINITY® ultrasound contrast agent or known hypersensitivity to perflutren microsphere or its components, e.g., polyethylene glycol. - Known sensitivity to gadolinium-based contrast agents
* Active seizure disorder or epilepsy (seizures despite medical treatment) for a minimum of 4 weeks prior to first cycle/Exablate BBBD procedure captured by history
* Patients with positive HIV status. - Immunosuppression (corticosteroids to prevent/treat brain edema are permitted)
* Cerebral or systemic vasculopathy, including intracranial thrombosis, vascular malformation, cerebral aneurysm, or vasculitis
* Hypertension per age
* History of a bleeding disorder, coagulopathy or with a history of spontaneous tumour hemorrhage
* Anti-coagulant therapy, or medications known to increase risk of hemorrhage, (e.g., ASA, non-steroidal anti-inflammatory drugs [NSAIDs], statins) within washout period prior to treatment
* Patient receiving bevacizumab (Avastin) therapy or increasing doses of steroids
* Symptoms and signs of increased intracranial pressure
* Previous participation in other chemotherapy, molecularly targeted therapy or immunotherapy treatment-related phase 1 or 2 trials
* Tumor not visible on any pre-therapy or post-radiation imaging

Ages: 5 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 10 (Estimated)
Dates: Start 2023-01-04 (Actual); Primary Completion 2026-01 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Adverse Events | 2 years
  All adverse events from first treatment to end of study will be documented and reported according to the CTCAE terminology and severity scale

SECONDARY OUTCOMES:
Blood Brain Barrier Disruption (BBBD) | Immediately post BBBD sonication
  BBBD will be assessed as a comparative ratio measured in pre and post-sonication contrast-enhanced MR images

OTHER OUTCOMES:
Tumor Volume | Immediately post BBBD sonication
  Average volume of contrast-enhancement on post sonicated MRI scans will be compared with pre-sonicated scans
Progression Free Survival (PFS) and Overall Survival (OS) | 2 years
  PFS will be assessed based on the Response Assessment in Pediatric Neuro-Oncology (RAPNO) scale. Tumor related biomarkers will be compared before and after the BBBD procedure

CONTACTS AND LOCATIONS:
Locations (1):
- Sunnybrook Research Institute, Toronto, Ontario, Canada